CLINICAL TRIAL: NCT05657652
Title: Venetoclax, Cladribine Plus Low-dose Cytarabine for Relapsed/Refractory Philadelphia Chromosome-negative (Ph-) B-cell Acute Lymphoblastic Leukemia (B-ALL): a Single-arm, Multicenter Study
Brief Title: CAV Regimen for R/R Ph- B-ALL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Jining Medical University (Other); The Second People's Hospital of Huai'an (Other); The First Affiliated Hospital of Bengbu Medical University (Other); Northern Jiangsu People's Hospital (Other); Affiliated Hospital of Nantong University (Other); Suzhou Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Sheng-Li Xue, MD, Professor, The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZBALL01
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: venetoclax; cladribine; cytarabine; relapsed/refractory ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence | interventions — Cladribine; Cytarabine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAV regimen (Experimental)
  Interventions: Drug: cladribine, cytarabine,venetoclax

INTERVENTIONS:
Drug: cladribine, cytarabine,venetoclax — Cladribine 5 mg/m2/day, cytarabine 20mg q12h, venetoclax 100mg d1, 200 d2, 400 mg/day from day 3 to day 21.

SUMMARY:
This study aims to investigate the efficacy and safety of cladribine, venetoclax combined with cytarabine and venetoclax (CAV regimen) for relapsed/refractory (R/R) Philadelphia Chromosome-negative (Ph-) B-cell acute lymphoblastic leukemia (B-ALL).

DETAILED DESCRIPTION:
Relapse is common in Ph- B-ALL and a proportion of patients present refractory to initial treatment. Treatments for these patients consist immunotherapy and conventional chemotherapy. The former is too expensive and the latter has a low remission rate. Treatment for R/R Ph- B-ALL still remains a challenge. The efficacy and safety of cladribine, venetoclax and cytarabine (CAV) has not been explored in ALL. Thus investigators design such a clinical trial to investigate the efficacy and safety of CAV regimen for R/R Ph- B-ALL.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 15-70 years old.
2. Patients diagnosed with R/R Ph- B-ALL.
3. Patients with ALL must meet one of the following criteria, A or B: A: Refractory ALL disease was defined as follows: (1) failure to attain CR following exposure to at least 1 courses of standard induction therapy; B: Relapsed ALL disease was defined as follows: (1) reappearance of leukemic blasts in the peripheral blood after CR; or (2) detection of ≥ 5% blasts in the BM not attributable to another cause (e.g., BM regeneration after consolidation therapy); or (3) extramedullary relapse.
4. ECOG performance status score less than 2.
5. Expected survival time ≥ 12 weeks.
6. Patients without serious heart, lung, liver, or kidney dysfunction.
7. Able to understand and provide informed consent.

Exclusion Criteria:

1. Patients who are allergic to the study drug or drugs with similar chemical structures.
2. Pregnant or lactating women, and women of childbearing age who do not want to practice effective methods of contraception.
3. Active infection.
4. Active bleeding.
5. Patients with new thrombosis, embolism, cerebral hemorrhage, or other diseases or a medical history within one year before enrollment.
6. Patients with mental disorders or other conditions.
7. Liver function abnormalities (total bilirubin > 1.5 times of the upper limit of the normal range, ALT/AST > 2.5 times of the upper limit of the normal range or patients with liver involvement whose ALT/AST > 1.5 times of the upper limit of the normal range), or renal dysfunction (Ccr<50ml/h).
8. Patients with a history of clinically significant QTc interval prolongation (male > 450 ms; female > 470 ms), ventricular heart tachycardia and atrial fibrillation, II-degree heart block, myocardial infarction attack within one year before enrollment, and congestive heart failure, and patients with coronary heart disease who have clinical symptoms and requiring drug treatment.
9. Surgery on the main organs within the past six weeks.
10. Drug abuse or long-term alcohol abuse that would affect the evaluation results.
11. Patients who have received organ transplants.
12. Patients not suitable for the study according to the investigator's assessment.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | ORR assessment is measured on days 21 from the start of CAV regimen
  The overall response (completed remission, completed remission with incomplete blood count recovery)

SECONDARY OUTCOMES:
Overall Survival (OS) | 2 years
  OS is measured from the time of enrollment to this trial to the date of death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive.
Progression-Free Survival (PFS) | 2 years
  PFS is measured from the time of enrollment to this study to progression or death.
Adverse events | 1 month
  It is evaluated and graded according to CTCAE 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China